CLINICAL TRIAL: NCT02016456
Title: An Evaluation of Transcranial Magnetic Stimulation in the National Health Service
Brief Title: TMS Treatment for Depression in the National Health Service
Acronym: TDEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mental Health Nottingham (Other)
Collaborators: Nottinghamshire Healthcare NHS Trust (Other Government)
Responsible Party: Principal Investigator, Sudheer Lankappa, Consultant Psychiatrist, Institute of Mental Health Nottingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMH/021213
Record Dates: First submitted 2013-12-15; First posted 2013-12-20 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Depression
Keywords: Transcranial Magnetic Stimulation; Neuronavigation; Magnetic Resonance Imaging
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Theta-Burst Stimulation (Experimental): Theta-Burst protocol for transcranial magnetic stimulation on dorsolateral prefrontal cortex (exact location to be determined using neuronavigation guided by Magnetic Resonance Imaging)
  Interventions: Device: Theta-Burst Stimulation
- High Frequency stimulation (Active Comparator): High frequency Transcranial Magnetic Stimulation using the standard protocol for depression, on left dorsolateral prefrontal cortex.
  Interventions: Device: High frequency stimulation

INTERVENTIONS:
Device: Theta-Burst Stimulation — At 80% motor threshold determined using single pulse stimuli. Depending on the hemisphere determined by connectivity analysis and neuronavigation in each individual, either continuous (left prefrontal) or intermittent (right prefrontal) train of pulses will be delivered.
  Arms: Theta-Burst Stimulation
Device: High frequency stimulation — Left prefrontal stimulation. 120% motor threshold with a pulse sequence of 10 Hz for 4 seconds, followed by a 26 second quiet period. Treatment will last for a total of 37.5 minutes this is a total of 3,000 pulses
  Arms: High Frequency stimulation

SUMMARY:
This research programme purports to test the effectiveness of two Transcranial Magnetic Stimulation (TMS) protocols (Repetitive high frequency protocol and Theta Burst protocol) in reducing the symptoms of depression. The study also uses Magnetic Resonance Imaging (MRI) scans to improve the localization of TMS targets.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of depressive disorder (DSM-IV)
* Diagnosis of treatment resistance (at least stage 1 as defined by Thase & Rush, 1997 for depression)
* Female or male between 18 and 70 years

Exclusion Criteria:

* History of Bipolar disorder
* Clinically relevant neurological comorbidity such as brain neoplasm, cerebral vascular events, epilepsy, neurodegenerative disorders, prior brain surgery
* Metal objects in and around body that cannot be removed
* Pregnancy
* Cardiac pacemaker or implanted medication pump
* Major unstable medical illness
* Change in prescribed medication in the 2 weeks preceding the start of TMS trial
* Current alcohol/stimulant dependence with propensity for toxic/withdrawal seizures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-10; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Proportion of responders defined as subjects with 50% reduction in the 17-item Hamilton Depression Scale Score | 4 weeks

SECONDARY OUTCOMES:
Mean change in Beck Depression Inventory scores | 4 weeks

OTHER OUTCOMES:
Change in processing speed (using modified digit-symbol test) scores | 4 weeks and 3 months
Change in Clinical Global Impression scores | 4 weeks and 3 months
Change in Social and Occupational Functioning Assessment scores | 4 weeks and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sudheer Lankappa, MRCPsych, Principal Investigator — Nottinghamshire Healthcare NHS Trust
Locations (1):
- Neuromodulation Unit, Nottinghamshire Healthcare NHS Trust, Nottingham, England, United Kingdom

REFERENCES:
- See also: Related Info — http://www.nlm.nih.gov/medlineplus/depression.html